CLINICAL TRIAL: NCT05698862
Title: Mapping the Impact of Gut Bacteria on Brain and Behaviour Through the Lens of GABA (GutBrainGABA)
Brief Title: Mapping the Impact of Gut Microbiota on Brain and Behavior Through the Lens of GABA
Acronym: GutBrainGABA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Bhismadev Chakrabarti, Professor of Neuroscience and Mental Health, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GBGABAWP2
Record Dates: First submitted 2023-01-03; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Gamma Amino Butyric Acid (GABA); Brain function; Gut microbiota; Behaviour; Probiotics
MeSH Terms: conditions — Behavior | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic supplement (Lactobacillus brevis)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo (maltodextrin)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants will be required to take a probiotic supplement of Lactobacillus brevis daily (1 capsule 5B CFU/day)
  Arms: Probiotic
Dietary Supplement: Placebo — Participants will be required to take the placebo maltodextrin daily (1 capsule/day)
  Arms: Placebo

SUMMARY:
Gut microbiota produce different metabolites within the human body, which include neurotransmitters. Animal studies have demonstrated a critical role for the gut microbiota in various aspects of brain and behavioural function, and a smaller number of studies in humans have shown differences of gut microbiota composition in psychiatric conditions. However, almost nothing is known about the impact of neurotransmitters produced by the gut microbiota on human brain and behaviour.

The way in which differences in brain, behaviour and personality traits are associated with the gut microbiota, and how they are influenced by a probiotic will be explored, with a special focus on GABA (Gamma Amino Butyric Acid).

Abnormalities of microbiota composition have been identified in metabolic disorders, such as inflammatory bowel disease and obesity, and psychiatric conditions, such as depression and anxiety.

The aim of this intervention trial will be to answer the following fundamental questions:

1. Does the population of gut bacteria capable of producing GABA modulate brain-based measures of GABA?
2. Does the population of gut bacteria capable of producing GABA influence performance in behavioural tasks known to depend on GABA-ergic function?

The impact of a GABA producing probiotic on the measures of GABA in the brain and serum, relevant metabolites in blood, faecal and urine samples and performance in GABA dependent behavioural tasks will be investigated in this trial.

DETAILED DESCRIPTION:
This interventional trial will involve a double-blind placebo-controlled crossover trial structured in 4 appointments: week 0 (W0), week 4 (W4), week 8 (W8) and week 12 (W12). The study will therefore last 12 weeks, and will include a screening visit and 4 study visits.

The interventional study has a cross-over design, and participants will therefore be invited to consume both the active probiotic supplement and the placebo at different times. The probiotic supplement (Lactobacillus brevis) was chosen based on the ability to produce GABA in vitro (Monteagudo et al., 2022). The placebo will be maltodextrin The products will be provided as capsules and are identical in texture and appearance.

For participants to be considered compliant and therefore included in the study they will be require:

1. to take the probiotic supplement or placebo at least 6 out of every 7 days of the trial for the week period;
2. to provide faecal, blood and urine samples and to be tested with a battery involving behaviour and brain measures relating to GABA levels/activity and
3. to complete a food diary using an online app once every 4 weeks.

As age and BMI are factors associated with significant variation in gut microbiota composition/brain and behaviour functioning, both study arms will be matched on these criteria.

All interested Individuals will be invited to complete an initial screening questionnaire, which includes questions related to a) the study inclusion criteria. Individuals who meet the study inclusion criteria will then be asked to complete b) an MRI contraindications questionnaire and, in absence of any MRI-related contraindications, they will be asked to c) complete a medical/lifestyle questionnaire to confirm the absence of any exclusion criteria.

Individuals who meet the inclusion criteria will be invited to attend a screening visit at the University of Reading for familiarisation with the procedures and for any clarification they might need. Participants will be provided with a sample collection kit (for faecal and urine sample collection), will be instructed on how to use it, and will be asked to track their diet using an online app (eNutri).

All study appointments will take place at the University of Reading. On the day of the study appointment, participants will be asked to provide a fresh faecal sample and spot urine sample (first morning urine), collected using the sample kit they were provided with at the screening visit. A venous blood sample (equal to 10ml/ 2tsp) will be collected by experienced and trained phlebotomists at the University of Reading. Participants will then undergo a neuroimaging battery, which will include structural magnetic resonance images, magnetic resonance spectroscopy (MRS) to quantify concentrations of GABA in determined regions of the brain, and functional magnetic resonance imaging to evaluate functional connectivity between brain areas. Participants will then complete a battery of GABA-dependent behavioural assays including a facial emotion recognition task, a motor learning task, and a tactile frequency discrimination task. Participants will then complete the Autism Spectrum Quotient (AQ), the State and Trait Anxiety Inventory (STAI), and the Centre for Epidemiological Studies Depression Scale (CES-D). Participants will complete this battery of tasks at each of the four study visits at W0, W4, W8 and W12.

At the end of visit 1 (W0), participants will be provided with either the probiotic OR placebo supplement to consume daily for the next 4 weeks, i.e. between study visits 1 and 2. At the end of visit 2 (W4), participants will not be provided with any supplements as they will enter their 4-week period of washout. At the end of visit 3 (W8), participants will be provided with either the probiotic OR placebo supplement to consume daily for the next 4 weeks. If the participant received the probiotic following visit 1, they will receive the placebo at this point, and vice versa. Participants will be asked to take this daily until their fourth and final study visit (W12). Study visit 4 finalises the study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Right-handed
* Caucasian/White
* Between 18 and 50 years of age
* Grew up in the UK or other European country
* Body Mass Index 18.5 to 30.

Exclusion Criteria:

* Use of antibiotics within the last 3 months
* Use of protonic pump inhibitors (PPIs) within the last 3 months
* Current or history of regular smoking within the last 6 months
* Regular consumption of >14 units of alcohol per week
* Current use of psychotropic drugs for medicinal or recreational purposes
* Current use of probiotic/prebiotic supplements
* Current diagnosis of neurological, developmental or psychiatric condition
* Current diagnosis of gut microbiota related conditions such as inflammatory bowel disease or irritable bowel syndrome

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in GABA concentrations in the brain assessed using Magnetic Resonance Spectroscopy (MRS) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Concentrations of GABA will be quantified using MRS. MRS data will be analysed separately in the time domain using an open-source magnetic resonance spectroscopy analysis tool, such as Osprey.
Changes in GABA-ergic activity in the sensorimotor component of the resting state network assessed using resting state functional Magnetic Resonance Imagine (rs-fMRI) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  GABA-ergic activity will be measured using rs-fMRI. MRI data will be analysed..
Changes in GABA concentrations in urine assessed by Liquid chromatography-mass spectrometry (LC-MS). | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Concentrations of GABA will be measured in urine samples by LC-MS.
Changes in GABA concentrations in serum assessed by Liquid chromatography-mass spectrometry (LC-MS). | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Concentrations of GABA will be measured in serum samples by LC-MS.

SECONDARY OUTCOMES:
Changes in faecal bacteria quantity assessed by Fluorescent In Situ Hybridisation Followed by Flow Cytometry (FISH-FCM) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Quantity of faecal bacteria will be assessed by FISH-FCM
Changes in compositional diversity of faecal microbiota attributable to intervention assessed by 16S ribosomal RNA (16S rRNA) gene amplicon sequencing | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment)
  Compositional diversity of faecal microbiota attributable to intervention will measured by 16S rRNA sequencing methods
Changes in metabolic profile in faecal samples assessed by Nuclear Magnetic Resonance spectroscopy (NMR) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  The metabolic profile will be measured in faecal samples using NMR
Changes in metabolic profile in urine samples assessed by Nuclear Magnetic Resonance spectroscopy (NMR) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  The metabolic profile will be measured in urine samples using NMR
Changes in metabolic profile in serum samples assessed by Nuclear Magnetic Resonance spectroscopy (NMR) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  The metabolic profile will be measured in serum samples using NMR
Changes in blood pressure assessed by measures of systolic and diastolic blood pressure | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Blood pressure will be recorded during the intervention using an upper arm blood pressure monitor
Changes in motor function performance assessed by reaction time | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Motor performance data will be calculated by averaging the reaction time from correct trials (i.e., where participants pressed the button corresponding to the visual sequence presented).
Changes in emotion recognition performance assessed by reaction time and accuracy | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Emotion recognition task accuracy and reaction time will be calculated in response to six emotions and a neutral facial expression.
Changes in tactile discrimination performance assessed by reaction time, static threshold and dynamic threshold | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Tactile discrimination reaction time and thresholds will be obtained from each participant using established 'staircase' threshold estimation procedures.
Changes in levels of trait and state anxiety assessed by the State-Trait Anxiety Inventory (STAI) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Trait and state levels of anxiety will be assessed by the STAI questionnaire
Changes in levels of depression assessed by the Centre for Epidemiological Studies Depression questionnaire (CES-D) | 1. Baseline (Week 0), 2. Following intervention (Week 4 or Week 12, depending on intervention arm assignment), 3. Following washout (Week 8), 4. Following placebo (Week 4 or Week 12, depending on intervention arm assignment)
  Levels of depression will be assessed by the CES-D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bhismadev Chakrabarti, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No